CLINICAL TRIAL: NCT06019286
Title: Novel Predictors of Premature Aging in COPD Patients: SCINEXA Score and Laboratory Markers
Brief Title: Novel Predictors of Premature Aging in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Refaat Mahmoud, principal investigator, Assiut University
Other Study IDs: premature aging in COPD
Record Dates: First submitted 2023-08-19; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: COPD
Keywords: premature aging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Aging, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD cases: COPD patients for whom biological marker and dermatological score will be measured
  Interventions: Diagnostic Test: SCINEXA score
- Control group: non COPD subjects for whom biological marker and dermatological score will be measured
  Interventions: Diagnostic Test: SCINEXA score

INTERVENTIONS:
Diagnostic Test: SCINEXA score — - 18 signs of extrinsic aging of SCINEXA score: sunburn, freckles, actinic lentigo, hyperpigmentation and/or melasma, change in phototype, yellowness, pseudoscars, coarse wrinkles, solar elastosis, cutis rhomboidalis, elastosis, comedones and cysts of Favre-Racouchot, xerosis, teleangectasias, permanent erythema, actinic keratosis, basal cell carcinoma, squamous cell carcinoma and malignant melanoma (extrinsic SCINEXA score). Each item will be scored as 0 (none), 1 (mild), 2 (moderate) or 3 (severe). For some items (uneven pigmentation, cutis rhomboidalis nuchae, elastosis, comedones and cysts of Favre Racouchot, and malignant skin tumors, a binary scale was used: (yes) or (no). Maximun possible score is 54
  Other Names: growth hormone level

SUMMARY:
•Examine whether COPD is associated with accelerated aging using a biological marker of aging and dermatological score

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) results from gene(G)-environment(E) interactions occurring over the lifetime(T) of the individual (GETomics) that can damage the lungs and/or alter their normal development/aging processes.

In COPD, processes including oxidant/antioxidant, protease/antiprotease, and proliferative/ antiproliferative balance, and the control of the inflammatory response become dysfunctional, as in aging. A close relationship between the pathogenesis of COPD and aging has been reviewed, and an increase regarding aging has been identified Aging is defined as a time-dependent progressive loss of physiological integrity, resulting in impaired function and increased vulnerability to death many chronic diseases are dependent on age and encompass physiological mechanisms related to the aging process The interconnection of the different markers of aging has not yet been studied in clinical subjects. We hypothesized that these markers, representing different interrelated aspects of the aging process, are altered in a cohort of COPD patients compared to the control group. These markers include growth hormone(GH), "Red cell distribution width (RDW) and SCINEXA (SCore for INtrinsic and EXtrinsic skin Aging) score as a read-out of biological age. SCINEXA is a validated score which measures the intrinsic and extrinsic factors regarding chronological skin aging and aging due to chronic exposure to ultraviolet (UV) radiation, Respectively.

The major feature of aging is the role of hormones as key regulators of human muscle metabolism and physical function. Growth hormone (GH) actions impact growth, metabolism, and body composition and have been associated with aging and Longevity. While, red cell distribution width (RDW), a part of the standard complete blood count (CBC), is a simple and non-invasive parameter that can be used as a biomarker in evaluating the severity and mortality rates in COPD patients in acute attacks. Also, Elevated RDW has been associated with degenerative conditions in aging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD attending outpatient are eligible for inclusion as cases. Control group is non COPD healthy controls.

Exclusion Criteria:

* • Patients refused to participate in the study.

  * Patients unable to perform the spirometry test.
  * Patients had a history of hormone disorder or malignant disease.
  * Patients received hormone replacement therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with COPD attending outpatient clinic either for follow up or newly diagnosed are eligible for inclusion as cases. Control group is non COPD healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
SCINEXA score in relation to COPD patient chronological age. | 1 week
  measuring SCINEXA score (Score for Intrinsic and Extrinsic skin Aging) in COPD patients and in control group and comparing it with chronological age. - 18 signs of extrinsic aging, each item will be scored as 0 (none), 1 (mild), 2 (moderate) or 3 (severe). For some items (uneven pigmentation, cutis rhomboidalis nuchae, elastosis, comedones and cysts of Favre Racouchot, and malignant skin tumors, a binary scale was used: (yes) or (no). Maximun possible score is 54
Level of GH and RDW in relation to COPD patient age. | 1 week
  measuring level of GH and in COPD patients and control group
Comparing level of GH with the chronological age | 1 week
  Compare level of GH with the chronological age of patients and controls to detected premature aging

CONTACTS AND LOCATIONS:
Overall Officials: Eman Fathy Ahmed, Dr., Study Chair — Assiut University; Heba Hassan Sayed, DR., Study Chair — Assiut University; Salma Mokhtar Osman, DR., Study Chair — Assiut University; Amal Adel Rayan, Dr., Study Chair — Assiut University

REFERENCES:
- [Background] Brat K, Svoboda M, Zatloukal J, Plutinsky M, Volakova E, Popelkova P, Novotna B, Dvorak T, Koblizek V. Prognostic Properties of the GOLD 2023 Classification System. Int J Chron Obstruct Pulmon Dis. 2023 Apr 20;18:661-667. doi: 10.2147/COPD.S410372. eCollection 2023. PMID 37114105
- [Background] Barnes PJ. Mechanisms of development of multimorbidity in the elderly. Eur Respir J. 2015 Mar;45(3):790-806. doi: 10.1183/09031936.00229714. Epub 2015 Jan 22. PMID 25614163
- [Background] Jiang Z, Han X, Wang Y, Hou T, Dong Y, Han X, Welmer AK, Launer LJ, Du Y, Qiu C. Red cell distribution width, anemia, and lower-extremity physical function among rural-dwelling older adults. Aging Clin Exp Res. 2022 Oct;34(10):2483-2491. doi: 10.1007/s40520-022-02187-9. Epub 2022 Aug 9. PMID 35943713
- [Background] Vierkotter A, Ranft U, Kramer U, Sugiri D, Reimann V, Krutmann J. The SCINEXA: a novel, validated score to simultaneously assess and differentiate between intrinsic and extrinsic skin ageing. J Dermatol Sci. 2009 Mar;53(3):207-11. doi: 10.1016/j.jdermsci.2008.10.001. Epub 2008 Dec 6. PMID 19059763